CLINICAL TRIAL: NCT07050550
Title: A Prospective Study of ¹⁸F-DFA PET Imaging for the Assessment of Liver Injury
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: The National Natural Science Foundation of China (NSFC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3.0
Record Dates: First submitted 2025-06-26; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Liver Injury
Keywords: liver injury; pet-ct; 18F-DFA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liver injury: liver injury

SUMMARY:
This study is a prospective exploratory clinical study aimed at evaluating the efficacy (sensitivity, specificity) of 18F-DFA PET imaging in assessing liver function damage. Subjects who meet the inclusion criteria are screened and enter this study to receive 18F-DFA PET imaging assessment, with clinical biochemical liver function indicators or liver puncture pathological examination as controls.

DETAILED DESCRIPTION:
Liver injury (LI) refers to a clinical syndrome caused by a rapid decline in liver function due to various causes in a short period of time, manifested by increased transaminase and bilirubin, pain in the liver area, abdominal distension, and jaundice. Acute treatment should be systematically carried out because liver injury can lead to liver dysfunction and even liver failure, and severe liver necrosis, which is life-threatening.

Currently, peripheral blood biochemistry, ultrasound, CT, MR, and liver biopsy are routinely used in clinical practice to evaluate the physiological and pathological changes of the liver during liver injury. The assessment of liver function from plasma is indirect, and marker molecules such as transaminases are diluted in the entire blood volume. During liver failure, when various processes such as inflammatory storms occur simultaneously, the results will be disturbed. Among the above methods, liver biopsy is the gold standard. However, liver biopsy only samples 1/50,000 to 1/100,000 of the liver, resulting in significant sampling errors. This heterogeneity of the liver is particularly significant when liver disease is heterogeneous, such as during liver injury and liver failure. Therefore, it is particularly important to find a non-invasive visualization that can display liver damage and liver failure in real time.

Vitamin C (VC), also known as L-ascorbic acid, is an essential water-soluble vitamin for the human body. As part of antioxidant and carbohydrate metabolism, VC participates in the circulation between liver cells and organs, mainly involving the hexuronic acid pathway, pentose phosphate cycle, glycolysis and gluconeogenesis. Glycogenolysis, as the main source of UDP-glucuronic acid, determines the rate of the hexuronic acid pathway leading to ascorbic acid synthesis. Glycogenolysis is regulated by oxidized and reduced glutathione. Therefore, glycogen, ascorbic acid and glutathione metabolism are interrelated, and the three together affect the antioxidant status of the liver. 6-Deoxy-6-[18F]fluoro-L-ascorbic acid (18F-DFA) is a radioactive tracer for positron emission tomography (PET) based on the structure of natural ascorbic acid (vitamin C). Recent literature reports show that 18F-DFA PET imaging can be used to evaluate liver damage and liver failure caused by acetaminophen. It can be seen that 18F-DFA PET molecular imaging is a promising diagnostic method for acute liver function injury, which may have higher sensitivity and specificity for the diagnosis of liver function injury and the evaluation of therapeutic efficacy.

In order to further observe the clinical diagnostic effect of this imaging method, we designed this prospective exploratory clinical study to further determine the effectiveness and safety of 18F-DFA PET imaging in evaluating liver function injury. Study purpose: To evaluate the efficacy (sensitivity, specificity) of 18F-DFA PET imaging in evaluating liver function injury with clinical biochemical liver function indicators or liver puncture pathological examination as control. To evaluate the correlation between liver uptake of 18F-DFA and liver function injury indicators (clinical biochemical liver function indicators or liver puncture pathological results).

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged between 18 and 80 years old; 2) Clinically diagnosed with liver damage (combined with medical history and laboratory tests, manifested as changes in liver enzymes, abnormal bilirubin metabolism, dysfunction of substance synthesis, and decreased biodegradation function, including indicators such as ALT, AST, ALP, GGT, albumin (Alb), TBil, and DBil); 3) Clinically diagnosed with liver failure (liver failure is a severe liver damage caused by multiple factors, resulting in severe dysfunction or decompensation of its synthesis, detoxification, excretion, and biotransformation functions, and a group of clinical syndromes with coagulation dysfunction, jaundice, hepatic encephalopathy, ascites, etc. as the main manifestations. Key points for the diagnosis of liver failure (a) Extreme fatigue, and severe gastrointestinal symptoms such as anorexia, vomiting, and abdominal distension; (b) Progressive deepening of jaundice (serum TBil ≥171μmol/L or daily increase ≥17.1μmol/L); (c) Bleeding tendency, plasma prothrombin activity (PTA≤40% or international normalized ratio (INR ≥ 1.5; (d) hepatic encephalopathy (grade II or above) or other complications.); 4) informed consent and able to accept follow-up, can understand and comply with the requirements of the study

Exclusion Criteria:

* 1) Patients with serious primary diseases of the heart, brain, kidney and hematopoietic system (i.e. Weber heart function grade D; hemoglobin (Hb) <10 g/dL, white blood cells (WBC) <3×109/L, platelets (PLT) <90×109/L; creatinine clearance (CrCl) <40 mL/min); 2) Patients with mental disorders or primary affective disorders; 3) Patients who cannot understand, follow the study protocol or sign the informed consent form; 4) Patients with contraindications to PET imaging (including pregnant women, breastfeeding women, women of childbearing age who have plans to have children in the near future, etc.); 5) Patients with allergies to imaging agents; 6) Patients who cannot cooperate with PET scanning due to hypoglycemia, severe pain or tremor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Clinical diagnosis of liver damage (combined with medical history and laboratory tests, manifested as changes in liver enzymes, abnormal bilirubin metabolism, dysfunction of substance synthesis and decreased biodegradation function, including indicators such as ALT, AST, ALP, GGT, albumin (Alb), TBil and DBil);
  2. Clinical diagnosis of liver failure (liver failure is a severe liver damage caused by multiple factors, resulting in severe dysfunction or decompensation of its synthesis, detoxification, excretion and biotransformation functions, and a group of clinical syndromes with coagulation dysfunction, jaundice, hepatic encephalopathy, ascites as the main manifestations. Key points for the diagnosis of liver failure (a) Extreme fatigue, and severe gastrointestinal symptoms such as obvious anorexia, vomiting and abdominal distension; (b) Progressive deepening of jaundice (serum TBil ≥171μmol/L or daily increase ≥17.1μmol/L); (c) Bleeding tendency, plasma prothrombin activity (PTA≤40
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the MAX%ID SUV in PET-CT imaging at 6 Months | The scan takes 10 minutes. After the scan is completed, patients will wait in the examination room for 1 hour before returning.
  Change from Baseline in the MAX%ID SUV in PET-CT imaging at 6 Months
To evaluate the correlation between liver uptake of 18F-DFA and liver function injury indicators (clinical biochemical liver function indicators or liver puncture pathological results). | The scan takes 10 minutes. After the scan is completed, patients will wait in the examination room for 1 hour before returning.
  To evaluate the correlation between liver uptake of 18F-DFA and liver function injury indicators (clinical biochemical liver function indicators or liver puncture pathological results).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowei XU, DOCTOR, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, we will compile all the data into an article and publish it, including the imaging and clinical data of all patients.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year after publication with no end date